CLINICAL TRIAL: NCT01171794
Title: Prevention of Altitude Illness With Non-steroidal Anti-inflammatory Study (PAINS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Grant S Lipman, PI, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SU-12012009-4443
Record Dates: First submitted 2010-07-27; First posted 2010-07-28 (Estimated); Results first posted 2017-04-20 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-11

CONDITIONS: Altitude Sickness
MeSH Terms: conditions — Altitude Sickness | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ibuprofen (Active Comparator): 600mg ibu TID
  Interventions: Drug: Ibuprofen
- placebo (Placebo Comparator): visually identical
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ibuprofen — 3 x 200mg (600mg total) x tid and one dosing on the subsequent day ( 4 doses total)
  Other Names: motrin
  Arms: ibuprofen
Drug: Placebo — identical number of visually identical tasteless pills as ibuprofen arm
  Arms: placebo

SUMMARY:
This is a research study on Altitude Illness. From the information collected and studied in this project we hope to learn more about Altitude Illness, including factors that may affect and prevent the development and progression of this condition. We hope to learn if the commonly used non-steroidal anti-inflammatory medication, ibuprofen can prevent altitude illness. Possible participants in this study are healthy adults who indicated they would like to participate, learn about altitude illness, and desire to hike Barcroft Peak. Stanford University researchers hope to enroll about 100 participants.

DETAILED DESCRIPTION:
This study was designed to bring together elements of prior studies and go one step further for definitive data on several points. The trial will employ two pharmaceutical intervention arms, which will compare placebo (the standard of care - information on prevention of altitude sickness) with the widely used NSAID ibuprofen. We will also determine Optic Nerve Sheath Diameter (ONSD) measurements via ultrasound in both the control and interventional arms. We will accomplish these objectives with a prospective, double blinded view of a large population of hikers who are ascending at their own rate in a true hiking environment: The White Mountain Research Station Owen Valley Lab (OVL) and Bancroft Station (BAR).

Primary hypothesis: Ibuprofen 600 mg TID will be superior to placebo in decreasing both the incidence and severity of AMS in high altitude travel.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Male or female volunteer
2. Age 18-65
3. Sea-level dwelling
4. Non pregnant
5. Have not been to high altitude in the past week
6. Can arrange for their own transportation to WMRS by friday evening the weekend of their study enrollment and are available the duration of the weekend of their study enrollment

Exclusion Criteria:

1. Age <18 or >65
2. Live at altitude > Sea Level +/- 1000'
3. Pregnant
4. Taking NSAIDs, Acetazolamide, or Corticosteroids
5. Allergic to NSAIDs or Aspirin, or have had adverse reaction to them in the past
6. Traveled or planning to travel to high altitude in the week prior to their enrollment.
7. Medical history of Brain Tumor, increased intercranial pressure, pseudotumor cerebri, ventricular shunts, loss of an eye, Asthma, HACE or HAPE.
8. Cannot arrange for their own transportation to WMRS or are unavailable for the duration of the weekend of their study enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2010-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grant S Lipman, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Result] Lipman GS, Kanaan NC, Holck PS, Constance BB, Gertsch JH; PAINS Group. Ibuprofen prevents altitude illness: a randomized controlled trial for prevention of altitude illness with nonsteroidal anti-inflammatories. Ann Emerg Med. 2012 Jun;59(6):484-90. doi: 10.1016/j.annemergmed.2012.01.019. Epub 2012 Mar 21. PMID 22440488

RESULTS

PARTICIPANT FLOW:
Groups:
- Ibuprofen: Ibuprofen : 3 x 200mg (600mg total) x tid and one dosing on the subsequent day ( 4 doses total)
- Placebo: Visually identical placebo
Period: Overall Study
Arm/Group | Ibuprofen | Placebo
Started | 47 | 42
Completed | 44 | 42
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Population: Participants meeting all inclusion criteria were analyzed
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibuprofen | Placebo | Total
Number analyzed (Participants) | 44 | 42 | 86
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 44 | 42 | 86
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.4 (14.5) | 34.2 (13.2) | 36.6 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 30 | 28 | 58

OUTCOME MEASURES:

1. Primary Outcome: Acute Mountain Sickness
Description: Lake Louise Criteria scores range from 0-15 with higher scores representing more severe symptoms; scores of 3 or greater with presence of a headache considered a positive diagnosis of acute mountain sickness
Time Frame: 2 days
Population: Participants meeting all inclusion criteria were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Ibuprofen | Placebo
Number analyzed (Participants) | 44 | 42
Participants | 19 | 26

2. Primary Outcome: Acute Mountain Sickness Severity
Description: Lake Louise Criteria scores range from 0-15 with higher scores representing more severe symptoms
Time Frame: 2 days
Population: Participants meeting all inclusion criteria were analyzed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ibuprofen | Placebo
Number analyzed (Participants) | 44 | 42
units on a scale | 3.2 (2.4) | 4.4 (2.6)

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Ibuprofen | Placebo
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/42
Other Adverse Events (participants affected / at risk) | 0/47 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes